CLINICAL TRIAL: NCT01793948
Title: A Double Blind Prospective Study of Metformin vs. Placebo in Overweight or Obese Post-menopausal Women at Elevated Risk for Breast Cancer
Brief Title: Metformin Hydrochloride vs. Placebo in Overweight or Obese Patients at Elevated Risk for Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anna Maria Storniolo (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Anna Maria Storniolo, Professor of Clinical Medicine, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IUCRO-0365; NCI-2013-00422 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1301010355 (Other: Indiana University IRB)
Record Dates: First submitted 2013-02-14; First posted 2013-02-18 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer; Obesity
MeSH Terms: conditions — Breast Neoplasms; Obesity | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (metformin hydrochloride) (Experimental): Patients receive metformin hydrochloride by mouth once daily on days 1-30 in course 1 and twice daily on days 1-30 thereafter. Treatment repeats every 30 days for 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: metformin hydrochloride; Other: laboratory biomarker analysis
- Arm II (placebo) (Placebo Comparator): Patients receive placebo by mouth once daily on days 1-30 in course 1 and twice daily on days 1-30 thereafter. Treatment repeats every 30 days for 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: placebo; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: metformin hydrochloride — Given PO
  Other Names: Glucophage
  Arms: Arm I (metformin hydrochloride)
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized clinical trial studies metformin hydrochloride in overweight or obese patients at elevated risk for breast cancer. Metformin hydrochloride may decrease the expression of early tumor makers in breast tissue of patients at increased risk for breast cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the changes in the signal pathway profiling of breast tissue using reverse phase proteomics in tissue biopsy of overweight or obese women at elevated risk for breast cancer treated with metformin (metformin hydrochloride) (850mg orally twice a day) for 12 cycles.

SECONDARY OBJECTIVES:

I. To determine the effect of metformin on breast tissue density of overweight or obese women at elevated risk for breast cancer using qualitative mammographic fat density criteria.

II. To determine the effect of metformin on the insulin axis in serum of overweight or obese women at elevated risk for breast cancer treated with metformin (850mg orally twice a day) for 12 cycles.

III. To determine the toxicities associated with metformin.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive metformin hydrochloride by mouth once daily on days 1-30 in course 1 and twice daily on days 1-30 thereafter. Treatment repeats every 30 days for 12 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive placebo by mouth once daily on days 1-30 in course 1 and twice daily on days 1-30 thereafter. Treatment repeats every 30 days for 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be post-menopausal women; post-menopausal women are defined as: (1) those >= 50 years of age who had not menstruated during the preceding 12 months or who had castrate follicle-stimulating hormone levels (> 40 IU/L), (2) those who had undergone a bilateral oophorectomy
* Patients must be at elevated risk for breast cancer based on strong family history or a history of breast biopsy documenting atypical hyperplasia anytime in the past; for this study strong family history is defined as having:

  * 1 first-degree (parent, offspring, sibling) relative =< 50 years old when diagnosed with breast cancer, or
  * >= 2 first-degree relatives of any age when diagnosed with breast cancer, or
  * >= 2 second-degree (aunts, uncles, grandparents, grandchildren, nieces, nephews, or half-siblings) maternal or paternal relatives diagnosed with breast cancer and at least 1 diagnosed at =< 50 years of age
* Patients must have a body mass index (BMI) >= 25.0 as calculated by the formula: weight in pounds / height squared x 703 = BMI; a BMI of:

  * 18.5-24.9 is considered normal;
  * 25.0-29.9 is considered overweight;
  * 30.0+ is regarded as obese
* Patients must be willing to complete a bilateral mammogram at baseline with repeat exam after 12 cycles of protocol therapy; patients who have had a mammogram within 1 month prior to registration to protocol therapy will not need to repeat the exam
* Patients must be willing to provide a core tissue biopsy at baseline and with repeat tissue collection after 12 cycles of protocol therapy
* White blood cell (WBC) >= 3.0 x 109/L
* Granulocytes (polymorphs + bands) >= 1.5 x 109/L
* Platelets >= 100 x 109/L
* Hemoglobin >= 110 g/L
* Aspartate aminotransferase (AST) =< 1.8 X upper limit of normal (ULN)
* Alanine aminotransferase (ALT) =< 1.8 X ULN
* Alkaline phosphatase =< 2 X ULN
* Serum creatinine =< 115 umol/L (1.3mg/dL)
* Serum bilirubin =< institution ULN (except for subjects with Gilbert's Disease who are eligible despite elevated serum bilirubin level)
* 12 hour fasting glucose level < 7.0 mmol/L
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1 within 28 days of registration
* Life expectancy of >= 5 years
* Subjects must be accessible for treatment, adverse event tracking and follow-up as determined by the treating physician
* Subject consent and authorization for the release of health information must be obtained according to local institutional guidelines

Exclusion Criteria:

* No history of any malignancy except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for >= 5 years
* No known diabetes (type 1 or 2) or baseline fasting glucose >= 7.0 mmol/L
* No known hypersensitivity or intolerance to metformin
* No condition associated with increased risk of metformin-associated lactic acidosis (e.g. congestive heart failure defined as New York Heart Association [NYHA] class III or IV functional status, history of acidosis of any type; habitual intake of 3 or more alcoholic beverages per day)
* No current treatment with metformin, sulfonylureas, thiazolidinediones or insulin for any reason
* No breastfeeding
* No concurrent or planned participation in randomized trials of weight loss or exercise interventions or trials targeting insulin, insulin-like growth factor 1 (IGF-1) or their receptors

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-04-16 (Actual); Primary Completion 2018-01-09 (Actual); Study Completion 2018-01-09 (Actual)

PRIMARY OUTCOMES:
Changes in the phosphorylation of proteins after metformin exposure | Baseline and 12 months
  Reverse phase proteomic assays (RPPA) will be performed to measure changes in the phosphorylation of proteins after metformin exposure. Changes in the phosphorylation of proteins after metformin exposure will be calculated and compared using two-sample t-tests. As a supplemental analysis, analysis of covariance (ANCOVA) will be used to model the 12 month levels adjusted for baseline. Assumptions for analysis will be checked and non-parametric methods used if needed; however it is expected that the data will be normally distributed on the log scale.

SECONDARY OUTCOMES:
Changes in ordinal level of breast density | Baseline and 12 months
  Changes in ordinal level of breast density will be performed using the breast density criteria previously established by Boyd and colleagues (New England Journal of Medicine 2007). Each image will be grouped into one of six categories: 0%, <10%, 10-25%, 25-50%, 50-75% and >75%. Changes will be compared between the two groups using Wilcoxon Rank-Sum tests.
Proportion of patients experiencing adverse events assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 30 days
  Will be tabulated by arm and grade.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria Storniolo, MD, Principal Investigator — Indiana University Melvin and Bren Simon Cancer Center
Locations (1):
- Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana, United States